CLINICAL TRIAL: NCT06163170
Title: Real-World Evaluation of Patient Characteristics, Treatment Patterns, Safety, and Efficacy of Nivolumab Monotherapy and Nivolumab in Combination With Ipilimumab for Pediatric Melanoma
Brief Title: A Study to Evaluate Treatment With Nivolumab Alone and Nivolumab Combined With Ipilimumab in Children With Melanoma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1068
Record Dates: First submitted 2023-10-20; First posted 2023-12-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with nivolumab +/- ipilimumab for unresectable/metastatic melanoma
  Interventions: Drug: Nivolumab +/- ipilimumab
- Participants treated with nivolumab as adjuvant therapy for resected stage IIB-IV melanoma
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab +/- ipilimumab — Participants treated with nivolumab +/- ipilimumab for unresectable/metastatic melanoma
  Groups: Participants treated with nivolumab +/- ipilimumab for unresectable/metastatic melanoma
Drug: Nivolumab — Participants treated with nivolumab as adjuvant therapy for resected stage IIB-IV melanoma
  Groups: Participants treated with nivolumab as adjuvant therapy for resected stage IIB-IV melanoma

SUMMARY:
The purpose of this study is to describe real-world safety outcomes in children with melanoma who are treated with nivolumab alone or nivolumab in combination with ipilimumab for unresectable or metastatic melanoma, or treated with adjuvant nivolumab after resection of stage IIB-IV melanoma. Demographic and clinical characteristics, and treatment patterns, will also be described in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed diagnosis of unresectable or metastatic cutaneous melanoma, or stage IIB-IV cutaneous melanoma who have undergone complete resection
* Initiated treatment with nivolumab monotherapy or in combination with ipilimumab for unresectable or metastatic melanoma, or as adjuvant therapy for resected stage IIb-IV melanoma, between January 1, 2015 and 6 months prior to data collection
* For the adjuvant nivolumab cohort, initiated treatment with nivolumab for stage IIb-IV melanoma within 12 weeks following index resection
* Aged <18 years at the time of nivolumab/ipilimumab treatment initiation
* At least 6 months of follow-up from index treatment date (unless deceased prior to end of 6 months)

Exclusion Criteria:

* Prior malignancy active within 3 years prior to nivolumab or ipilimumab treatment index date except for locally curable cancers that have been apparently cured (such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast)
* Receiving nivolumab therapy (monotherapy, combination with ipilimumab, or adjuvant therapy) for melanoma as part of a clinical trial during the study period

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric participants (<18 years of age) who were treated with nivolumab monotherapy or nivolumab combined with ipilimumab for unresectable or metastatic melanoma or treated with adjuvant nivolumab after resection of stage IIb-IV melanoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 100 days after treatment discontinuation
Incidence of all-cause adverse events | Up to 100 days after treatment discontinuation

SECONDARY OUTCOMES:
Participant year of birth | Six months prior to index date
Participant gender | Six months prior to index date
Participant race | Six months prior to index date
Participant ethnicity | Six months prior to index date
Participant state/region of residence | Six months prior to index date
Participant primary insurance payer at treatment initiation | Six months prior to index date
Date of initial melanoma diagnosis | Six months prior to index date
Date of index resection for participants treated with adjuvant nivolumab | Six months prior to index date
Participant height | Initiation of index treatment
Participant weight | Initiation of index treatment
Stage of melanoma at diagnosis, assessed by American Joint Committee on Cancer criteria | Six months prior to index date
Margins at index resection for participants treated with adjuvant nivolumab after resection | Six months prior to index date
Lymph node biopsy results | Six months prior to index date
Lymph node involvement - Stage III/IV only | Six months prior to index date
Tumor ulceration status | Six months prior to index date
Tumor ulceration characteristics | Six months prior to index date
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) | Initiation of index treatment
Lactate dehydrogenase level | Initiation of index treatment
Index treatment | Initiation of index treatment
Number of lines of therapy received for unresectable/metastatic melanoma | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Number of lines of therapy received post resection | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Disease response characteristics | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Disease recurrence characteristics | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Duration of therapy (DOT) | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Time to next treatment (TTNT) | From index therapy initiation to next subsequent systemic melanoma treatment post-nivolumab, death, or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Treatment-free interval (TFI) | From discontinuation of index treatment to date of initiation of subsequent therapy, assessed up to 108 months
Overall survival (OS) | From index therapy initiation to death or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Healthcare resource utilization assessed by the number of inpatient hospitalizations | From initiation of therapy until end of data collection date or death, whichever came first, assessed up to 108 months
Healthcare resource utilization assessed by the number of emergency department (ED) visits | From initiation of therapy until end of data collection date or death, whichever came first, assessed up to 108 months
Overall response rate (ORR) in participants with unresectable or metastatic disease | From index therapy initiation to the date of last follow-up/study end date, whichever came first, assessed up to 108 months
  Number of participants with complete or partial response divided by the total number of participants
Progression-free survival (PFS) in participants with unresectable or metastatic disease | From index therapy initiation to date of first documented disease progression, death, or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Time to initial response (TTR) in participants with unresectable or metastatic disease | From index therapy initiation to date of the first physician-reported response (complete or partial response), assessed up to 108 months
Duration of response (DOR) in participants with unresectable or metastatic disease | From date of first physician-reported response (complete or partial response) to date of the first physician-reported disease progression, death, or date of last follow-up/study end date, whichever came first, assessed up to 108 months
Time to progression (TTP) in participants with unresectable or metastatic disease | From index therapy initiation to date of physician-reported disease progression, or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Time to local disease recurrence in participants with resected disease | From index therapy initiation to date of last follow-up/study end date, whichever came first, assessed up to 108 months
Recurrence free survival (RFS) in participants with resected disease | From index therapy initiation to date of first melanoma recurrence, death, or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Time to distant metastases in participants with resected disease | From index therapy initiation to date of last follow/up or study end date, whichever came first, assessed up to 108 months
Distant-metastasis free survival (DMFS) in participants with resected disease | From index therapy initiation to date of first distant melanoma metastasis, death, or the date of last follow-up/study end date, whichever came first, assessed up to 108 months
Type of disease recurrence/metastasis in participants with resected disease | From index therapy initiation to date of last follow-up visit or study end date, whichever came first, assessed up to 108 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cardinal Health, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts